CLINICAL TRIAL: NCT03913494
Title: Transoral Daytime Neuromuscular Electrical Stimulation in Patients With Simple Snoring
Acronym: SnooZeal-snore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Associate Physician, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 181359
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea; Sleep; Snoring
Keywords: Upper Airway Conditioning; Snoring; Snore; Sleep; OSA; Sleep Apnea; Neurostimulation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4 Week Snoozeal Use (Experimental): Participants will take the device home and be required to use it for 20 minutes morning and night every day for at least 4 weeks. The SnooZeal records usage time to allow assessment of compliance.
  Interventions: Device: Transoral Neurostimulation Device (Snoozeal)

INTERVENTIONS:
Device: Transoral Neurostimulation Device (Snoozeal) — Use of the Transoral Neurostimulation Device for 20 minutes, morning and night, every day for at least 4 weeks.

SUMMARY:
Sleep Disordered Breathing (SDB) is a spectrum of conditions spanning from Simple Snoring to Severe Sleep apnea. SDB has multiple underlying mechanisms. Some portion of patients have issues with upper airway dilator muscle control; and such patients may be amenable to upper airway muscle training exercises using neuromuscular stimulation techniques. The investigators and others have published on the topic of neuromyopathy in the upper airway, defining a subgroup of OSA patients who may be amenable to training exercises. Based on this background, the investigators seek to test the hypothesis that upper airway tongue muscle training using transoral surface neuromuscular electrical stimulation may have benefits to patients with Simple Snoring.

ELIGIBILITY:
Inclusion Criteria:

• Confirmation of snoring: must have a live-in bed partner that reports ≥ 6 months history of habitual snoring (i.e. > 5 days per week)

Exclusion Criteria:

* AHI > 15/hr
* BMI > 35
* Non-English speakers (due to necessity to complete questionnaires)
* Inability to complete daily neuromuscular stimulation
* Other sleep disorders
* Tongue or lip piercing
* Pacemaker of implanted medical electrical devices
* Current or recent (within last 6 months) treatment for snoring or sleep apnea
* Previous oral or pharyngeal surgery other than dental
* Craniofacial skeletal or muscular abnormalities
* History of driving or other accidents due to sleepiness or an Epworth score (ESS)> 18
* Pregnant
* Cardiac (other than hypertension), pulmonary, renal, neurologic, neuromuscular or hepatic disease
* Medications with sedative or myorelaxant properties or effects on cardiac or pulmonary function
* Substantial alcohol (>3oz/day) or use of illicit drugs
* Psychiatric disorders (other than depression or anxiety)
* Snoring less than 20% of total sleep time during baseline polysomnography

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
NREM EMGgg | 6 hours
  Genioglossal muscle activity as measured by two 25 gauge needles each containing a Teflon-coated stainless steel recording wire (<0.1 mm in diameter with ~1 mm at the tip bared of Teflon and bent to form a small hook) placed perorally 1.5-2 cm into the body of the genioglossus muscle.
Change in percent total sleep time spent snoring | 6 hours
  Time spent snoring divided by total sleep time as determined by Polysomnogram

SECONDARY OUTCOMES:
Sleep Quality | 10 minutes
  A self-report questionnaire, titled the Pittsburgh Quality of Sleep Questionnaire (PSQI), asking several questions to determine quality of sleep over the past 1 month that will be scored and added together on a scale of 0-21.
Daytime Sleepiness | 10 minutes
  A self-report questionnaire, titled the Epworth Sleepiness Scale (ESS), asking subjects to rate their probability of falling asleep during different situations on a scale of 0-3. Scores are added together to determine how sleepy the subject feels during the day on a scale of 0-24

CONTACTS AND LOCATIONS:
Overall Officials: Robert Owens, MD, Principal Investigator — UCSD
Locations (2):
- United States (2):
  - Altman Clinical and Translational Research Institute, San Diego, California
  - University of California San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camacho M, Certal V, Abdullatif J, Zaghi S, Ruoff CM, Capasso R, Kushida CA. Myofunctional Therapy to Treat Obstructive Sleep Apnea: A Systematic Review and Meta-analysis. Sleep. 2015 May 1;38(5):669-75. doi: 10.5665/sleep.4652. PMID 25348130
- [Background] Camacho M, Guilleminault C, Wei JM, Song SA, Noller MW, Reckley LK, Fernandez-Salvador C, Zaghi S. Oropharyngeal and tongue exercises (myofunctional therapy) for snoring: a systematic review and meta-analysis. Eur Arch Otorhinolaryngol. 2018 Apr;275(4):849-855. doi: 10.1007/s00405-017-4848-5. Epub 2017 Dec 23. PMID 29275425
- [Background] Deary V, Ellis JG, Wilson JA, Coulter C, Barclay NL. Simple snoring: not quite so simple after all? Sleep Med Rev. 2014 Dec;18(6):453-62. doi: 10.1016/j.smrv.2014.04.006. Epub 2014 May 9. PMID 24888523
- [Background] Young T, Finn L, Hla KM, Morgan B, Palta M. Snoring as part of a dose-response relationship between sleep-disordered breathing and blood pressure. Sleep. 1996 Dec;19(10 Suppl):S202-5. doi: 10.1093/sleep/19.suppl_10.s202. PMID 9085511
- [Background] Wessolleck E, Bernd E, Dockter S, Lang S, Sama A, Stuck BA. Intraoral electrical muscle stimulation in the treatment of snoring. Somnologie (Berl). 2018;22(Suppl 2):47-52. doi: 10.1007/s11818-018-0179-z. Epub 2018 Sep 6. PMID 30595662